CLINICAL TRIAL: NCT02811432
Title: The OMWaNA Study: Operationalising Kangaroo Mother Care Before Stabilisation Amongst Low Birth Weight Neonates in Africa: a Multi-site Randomised Controlled Trial to Examine Mortality Impact in Uganda
Brief Title: Kangaroo Mother Care Before Stabilisation Amongst Low Birth Weight Neonates in Africa
Acronym: OMWaNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: MRC/UVRI and LSHTM Uganda Research Unit (Other); Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2023-09

CONDITIONS: Kangaroo Mother Care; Preterm Infant; Death; Neonatal; Hypothermia, Newborn
Keywords: Kangaroo mother care; Preterm; Low birthweight; Neonatal; Newborn; Randomised trial
MeSH Terms: conditions — Premature Birth; Perinatal Death; Hypothermia | interventions — Kangaroo-Mother Care Method; Standard of Care

STUDY DESIGN:
Masking Description: Masking of parents, caregivers, or healthcare workers was not possible due to the nature of the KMC intervention. The independent statistician who conducted the analyses was masked to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kangaroo mother care (Experimental): Skin-to-skin care initiated as soon as possible following randomisation
  Interventions: Other: Kangaroo mother care
- Standard care (Active Comparator): Incubator or radiant warmer
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Kangaroo mother care — Skin-to-skin care (target: at least 18 hours per day)
  Other Names: Skin-to-skin care
  Arms: Kangaroo mother care
Other: Standard care — Incubator or radiant warmer until neonate meets stability criteria; once stable (WHO indication for KMC certain), the baby can transition to routine (intermittent) KMC
  Arms: Standard care

SUMMARY:
We will conduct an individually randomised, controlled, superiority trial with two parallel groups; an intervention arm allocated to receive KMC and a control arm receiving 'standard' care. The primary aim is to examine the impact of KMC initiated before stabilisation on mortality within 7 days relative to standard care amongst neonates ≤2000g at four hospitals in Uganda. We hypothesise that neonates in the arm allocated to receive KMC before stabilisation will have a 25% overall reduction in mortality within 7 days compared to neonates allocated to receive standard care.

DETAILED DESCRIPTION:
METHODS Study setting, design, and participants The OMWaNA trial was an individually randomised, controlled, superiority trial with two parallel arms allocated in a 1:1 ratio to receive KMC initiated before stabilisation (intervention) or standard care (control). The trial was conducted in the neonatal units (WHO level-2) of five government hospitals in Uganda (appendix p 5). Infrastructure and equipment improvements as well as training were required prior to trial initiation, as described previously.10 All hospitals were provided with essential equipment and supplies to support the provision of KMC and level-2 newborn care. Details regarding study context and methods have been published in the trial protocol9 and are briefly summarised here. Ugandan practice is that maternity and newborn care should be provided free of charge in government health facilities;11 however, families are expected to support caregivers to meet essential needs such as meals.

The trial is reported here in accordance with the CONSORT guidelines. All live-born neonates, aged 1 to <48 hours and weighing 700-2000g, who were admitted to participating hospitals and for whom the indication for KMC was "uncertain" according to WHO guidance concerning clinical stability, defined as receiving ≥1 therapy (oxygen, continuous positive airway pressure [CPAP] where available, intravenous [IV] fluids, therapeutic antibiotics, anti-seizure medication), were eligible for inclusion. Exclusion criteria included triplet or higher multi-fetal pregnancy (unless pregnancy resulted in demise of ≥1 fetus) and parent/caregiver being unable/unwilling to provide either consent, KMC, and/or attend follow-up visits. Neonates with life-threatening instability, severe jaundice requiring immediate management, active seizures, or major congenital malformations were also excluded. The study was approved by the Research Ethics Committees of Uganda Virus Research Institute (GC/127/19/06/717), Uganda National Council of Science and Technology (HS 2645), and London School of Hygiene & Tropical Medicine (LSHTM, 16972). The trial was overseen by a steering committee and an independent data and safety monitoring board (DSMB).

Screening and informed consent All admitted neonates weighing ≤2000g were screened for eligibility by study staff. Stable neonates (meeting WHO 2019 criteria for KMC eligibility) were excluded and remaining neonates were assessed for eligibility. Those who met criteria for 'life-threatening instability' or who had conditions precluding KMC (e.g., seizures, jaundice), were reassessed every 3 hours up to 48 hours, after which they were excluded. Written informed parental consent was obtained for all participants.

Randomisation, allocation concealment and masking A random allocation sequence was computer-generated using permuted blocks of varying sizes stratified by birthweight (<1000g, 1000-1499g, ≥1500g) and recruitment site. Allocation concealment was done by programming the allocation sequence into the screening database and revealing treatment group only when screening of eligible neonates was complete. Neonates from multiple births (twins or triplets) were allocated to the same arm according to first-born allocation.14 Masking of parents, caregivers, or healthcare workers was not possible due to the nature of the KMC intervention.

Procedures In the intervention arm, KMC was initiated soon after randomisation. Neonates were naked except for hat and diaper, placed prone and skin-to-skin on caregiver's chest, and secured using a KMC wrap. Adjustable beds were provided to facilitate continuous skin-to-skin care. KMC duration was charted by caregivers and verified by study staff. When not in KMC (e.g., during maternal bathing), incubator or radiant heater care was commenced. Study personnel, in addition to hospital staff, provided continuous KMC counselling throughout the hospitalisation. Control arm neonates were cared for in an incubator or radiant heater, as per hospital practice. Caregivers could have physical contact with their newborn but skin-to-skin contact was not initiated until stability criteria were met.9 Once stable, newborns were transferred to routine (intermittent) KMC. Neonates in both arms received standard clinical care according to hospital guidelines.

ELIGIBILITY:
Inclusion criteria

* Liveborn at Jinja Hospital, Masaka Hospital, Entebbe Hospital, or Iganga Hospital
* Singleton or twin pregnancy
* Birthweight ≥700g and ≤2000g
* Chronological age 1-48 hours at time of screening
* Alive at time of recruitment
* Parent/caregiver able and willing to provide KMC
* Parent/caregiver willing to attend follow-up visit
* Indication for KMC "uncertain" according to WHO guideline concerning clinical stability: pragmatically defined as receiving ≥1 therapy: oxygen, CPAP, IV fluids, therapeutic antibiotics, phenobarbital

Exclusion criteria

* Outborn
* Result of triplet or higher order multifetal pregnancy
* Indication for KMC "certain" according to WHO guidelines: pragmatically defined as clinically well neonates receiving none of the above therapy-based criteria
* Severely life-threatening instability defined as SpO2 <88% in oxygen AND ≥1 of:

  * Respiratory rate <20 or >100 breaths/min
  * Apnoea requiring bag-mask ventilation
  * HR <100 or >200 bpm
* Severe jaundice requiring immediate management
* Active neonatal seizures
* Major congenital malformation
* Parent does not provide written informed consent to participate in trial
* Mother or neonate enrolled in another MRC/UVRI research project

Ages: 1 Hour to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2221 (Actual)
Dates: Start 2019-10-13 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joy E. Lawn, BMBS MPH PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (4):
- Uganda (4):
  - Entebbe, Entebbe
  - Iganga District Hospital, Iganga
  - Jinja Regional Referral Hospital, Jinja
  - Masaka Regional Referral Hospital, Masaka

IPD SHARING:
Plan to Share IPD: Yes
LSHTM Data Compass
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When main results paper is published - currently under review
Access Criteria: email to LSHTM data compass and agreement by study data sharing committee
URL: https://datacompass.lshtm.ac.uk/

REFERENCES:
- [Background] Medvedev MM, Tumukunde V, Mambule I, Tann CJ, Waiswa P, Canter RR, Hansen CH, Ekirapa-Kiracho E, Katumba K, Pitt C, Greco G, Brotherton H, Elbourne D, Seeley J, Nyirenda M, Allen E, Lawn JE. Operationalising kangaroo Mother care before stabilisation amongst low birth Weight Neonates in Africa (OMWaNA): protocol for a randomised controlled trial to examine mortality impact in Uganda. Trials. 2020 Jan 31;21(1):126. doi: 10.1186/s13063-019-4044-6. PMID 32005286
- [Background] Medvedev MM, Tumukunde V, Kirabo-Nagemi C, Greco G, Mambule I, Katumba K, Waiswa P, Tann CJ, Elbourne D, Allen E, Ekirapa-Kiracho E, Pitt C, Lawn JE. Process and costs for readiness to safely implement immediate kangaroo mother care: a mixed methods evaluation from the OMWaNA trial at five hospitals in Uganda. BMC Health Serv Res. 2023 Jun 10;23(1):613. doi: 10.1186/s12913-023-09624-z. PMID 37301974
- [Result] Tumukunde V, Medvedev MM, Tann CJ, Mambule I, Pitt C, Opondo C, Kakande A, Canter R, Haroon Y, Kirabo-Nagemi C, Abaasa A, Okot W, Katongole F, Ssenyonga R, Niombi N, Nanyunja C, Elbourne D, Greco G, Ekirapa-Kiracho E, Nyirenda M, Allen E, Waiswa P, Lawn JE; OMWaNA Collaborative Authorship Group. Effectiveness of kangaroo mother care before clinical stabilisation versus standard care among neonates at five hospitals in Uganda (OMWaNA): a parallel-group, individually randomised controlled trial and economic evaluation. Lancet. 2024 Jun 8;403(10443):2520-2532. doi: 10.1016/S0140-6736(24)00064-3. Epub 2024 May 13. PMID 38754454

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Skin-to-skin care initiated as soon as possible following randomisation
  Kangaroo mother care: Skin-to-skin care (target: at least 18 hours per day)
- Control: Incubator or radiant warmer
  Standard care: Incubator or radiant warmer until neonate meets stability criteria; once stable (WHO indication for KMC certain), the baby can transition to routine (intermittent) KMC
Period: Overall Study
Arm/Group | Intervention | Control
Started | 1110 | 1111
Completed | 1083 | 1102
Not Completed | 27 | 9

BASELINE CHARACTERISTICS:
Groups:
- Kangaroo Mother Care: Skin-to-skin care initiated as soon as possible following randomisation
  Kangaroo mother care: Skin-to-skin care (target: aiming for 18 hours per day)
- Total: Total of all reporting groups
Arm/Group | Kangaroo Mother Care | Standard Care | Total
Number analyzed (Participants) | 1110 | 1111 | 2221
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1110 | 1111 | 2221
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: hours] | 20.3 (11.6) | 21.5 (11.5) | 20.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 552 | 550 | 1102
  Male | 558 | 561 | 1119
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1110 | 1111 | 2221
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 1110 | 1111 | 2221

OUTCOME MEASURES:

1. Primary Outcome: Mortality Within 7 Days
Description: early neonatal mortality at 7 days
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1083 | 1102
Participants | 81 | 83

2. Secondary Outcome: Prevalence of Hypothermia at 24 Hours Post-randomisation
Description: Prevalence of hypothermia at 24 hours post-randomisation using axillary temperature was assessed using a digital thermometer.
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1096 | 1101
participants | 448 | 585

3. Secondary Outcome: Time From Intervention/Control Procedures Starting to Clinical Stabilisation
Description: Time-to-stabilization was defined as the first time at which a neonate had met all of the following criteria for a continuous period of at least 24 hours: breathing spontaneously with SpO2 >90% in room air; no need for supplemental oxygen or CPAP; respiratory rate 40-59 breaths per minute; no apneic episodes; heart rate 80-179 beats per minute; axillary temperature 36.0-37.4 °C; and no need for intravenous fluids.
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1081 | 1100
days | 5.1 [4.1 to 6.7] | 4.9 [3.8 to 6.5]

4. Secondary Outcome: Time From Starting Intervention/Control Procedures to Death
Description: The date and time of death were prospectively recorded from the death certificate for in-hospital deaths. For deaths occurring after discharge, the date was recorded based on parent/caregiver verbal report. Median and IQR of time-to-event calculated as the 50th and 25th to 75th percentile of the distribution of event times among those who experienced the event.
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Intervention | Control
Number analyzed (Participants) | 119 | 134
hours | 5.0 [2.5 to 10.7] | 5.9 [2.8 to 13.9]

5. Secondary Outcome: Mean Duration of Hospital Stay in Days
Description: The date and time of hospital admission and discharge were documented prospectively for the first admission episode.
Time Frame: 30 days
Population: at the 28-30 day visit
Measure: Mean (Standard Error); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1083 | 1102
days | 7.3 (0.15) | 6.1 (0.14)

6. Secondary Outcome: Proportion of Neonates Exclusively Breastmilk Feeding at Discharge
Description: Proportion of neonates who were exclusively breastmilk feeding at discharge, from the breast or by other means
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1083 | 1102
Participants | 959 | 978

7. Secondary Outcome: Mortality Within 28 Days
Description: All-cause mortality within 28 days. Vital status was documented at the 28-30-day follow-up visit. If participants did not attend, a telephone call was made the same day to ascertain outcome.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1051 | 1049
Participants | 119 | 134

8. Secondary Outcome: Frequency of Readmission
Description: Episodes in which a neonate was readmitted to the index hospital were prospectively recorded. Episodes in which a neonate was readmitted to a different hospital were recorded based on parent/caregiver verbal report.
Time Frame: 30 days
Population: by 28-30 day visit
Measure: Mean (Standard Error); unit: readmission count
Arm/Group | Intervention | Control
Number analyzed (Participants) | 848 | 840
readmission count | 0.02 (0.01) | 0.04 (0.01)

9. Secondary Outcome: Daily Weight Gain at 28 Days
Description: Mean daily weight gain was calculated as the difference between weight at enrollment and 28-30-day follow-up, as measured by the study scale.
Time Frame: 28 days
Population: by 28-30 day visit
Measure: Mean (Standard Error); unit: g/kg/day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 761 | 731
g/kg/day | 7.8 (0.3) | 7.1 (0.3)

10. Secondary Outcome: Infant-caregiver Attachment at 28 Days
Description: The intention-to-treat analysis assessed the mean difference in Maternal Infant Responsiveness Instrument score between the two arms. Scores range from 0 to 110, with higher scores indicating greater attachment.
Time Frame: 28 days
Population: day 28-30 visit
Measure: Mean (Standard Error); unit: MIRA score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 758 | 725
MIRA score | 85.4 (0.28) | 85.0 (0.28)

11. Secondary Outcome: Women's Well-being at 28 Days
Description: The intention-to-treat analysis assessed the mean difference in Women's Capabilities Index (WCI) score between the two arms. The WCI has a scale of 0 to 1, with higher scores indicating greater wellbeing. The analysis excluded duplicate entries for mothers of enrolled twins/triplets.
Time Frame: 28 days
Population: at the 28-30 day visit
Measure: Mean (Standard Error); unit: WCI score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 624 | 602
WCI score | 0.69 (0.01) | 0.68 (0.01)

ADVERSE EVENTS:
Time Frame: 28 days of age
Description: The site paediatrician was informed about SAEs within 24 h. SAEs were followed up by the site paediatrician until resolution, or until causality was determined as unrelated to the trial intervention. If an unexpected SAE occurred, potentially related to the trial intervention, a report was submitted to the Research Ethics Committees (REC) at UVRI and LSHTM within 48h, with a follow-up report provided. All SAEs were reported to Sponsor and DSMB as part of their respective reports.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 119/1051 | 134/1049
Serious Adverse Events (participants affected / at risk) | 124/1051 | 125/1049
Other Adverse Events (participants affected / at risk) | 180/1051 | 90/1049
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=1051) | Control (N=1049)
SAEs and other adverse events (Blood and lymphatic system disorders) | 8 (8) | 10 (10)
SAEs and other adverse events (Cardiac disorders) | 0 (0) | 1 (1)
SAEs and other adverse events (Gastrointestinal disorders) | 12 (12) | 7 (7)
SAEs and other adverse events (Respiratory, thoracic and mediastinal disorders) | 59 (59) | 63 (63)
Neonatal jaundice (Hepatobiliary disorders) | 4 (4) | 6 (6) — Neonatal jaundice with elevated bilrubin
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) — Acute kidney injury with elevated creatinine
Neurological disorders (Nervous system disorders) | 8 (8) | 9 (9) — Neurological disorders including seizures, intracranial haemorrhage
neonatal infections (Infections and infestations) | 34 (34) | 35 (35) — Sepsis suspected or confirmed
Hyperthermia (General disorders) | 0 (0) | 2 (2) — Hyperthermia
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=1051) | Control (N=1049)
Neonatal jaundice (Hepatobiliary disorders) | 180 (180) | 90 (90) — Neonatal jaundice

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT02811432/Prot_001.pdf
  • Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT02811432/SAP_002.pdf